CLINICAL TRIAL: NCT01369563
Title: Non-interventional Clinical Trial, to Assess the Efficacy, Safety and Tolerability of Ciclesonide 200 Mcg Once Daily, Applied as a Nasal Spray for Four Weeks, in the Treatment of Intermittent and Persistent Rhinitis
Brief Title: Efficacy, Safety & Tolerability of Ciclesonide 200mcg Spray 4 Weeks Treatment for Intermittent & Persistent Rhinitis
Acronym: SISRIP
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: MX028; U1111-1133-6326 (Registry Identifier: WHO)
Record Dates: First submitted 2011-06-07; First posted 2011-06-09 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-09

CONDITIONS: Perennial Rhinitis; Seasonal Rhinitis
Keywords: rhinitis; ciclesonide; intermittent rhinitis; persistent rhinitis
MeSH Terms: conditions — Rhinitis

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
To assess the efficacy, safety and tolerability of ciclesonide 200 mcg once daily, applied as a nasal spray for four weeks. The main outcome will be the improvement on global and individual typical and associated symptoms of intermittent or persistent rhinitis.

DETAILED DESCRIPTION:
Study design:

This is a prospective national wide Non- Interventional study. Patients number 2400 CRFs will be distributed in order to obtain a ITT (Intention to Treat) sample of 1800 (75%) patients, and PP (Per Protocol) sample of 1100 patients (60%).

400 patients will be applied to "prick test" and the results will be analyzed to determine the prevalence and response to treatment according to the diagnosis of allergic rhinitis.

Eligible population Male or female external patients over 18 years and under 50 years with active rhinitis (anterior or posterior rhinorrhea, sneezing, nasal congestion and itching) persistent (≥ 4 days a week for 4 consecutive weeks) or intermittent (< 4 days a week for ≤ 4 consecutive weeks), with medical history of rhinitis 2 years prior to their participation in this study and whose nasal symptoms have been severe enough to require continuous or intermittent treatment (it requires a patient's symptoms need treatment at least for a 4 weeks period). All patients have to sign the informed consent or give verbal confirmation prior to their inclusion in the study.

Evaluation criteria:

Primary:

Symptoms relief of intermittent or persistent rhinitis .

Secondary:

Safety profile (MedDRA adverse events), tolerability and treatment compliance.

Collective evaluation:

The PP population will be considered for confirmatory analysis. The key variable "symptom relief" will be assessed for the Intent-to-treat population or ITT for comparison.

Statistical analysis:

The investigators will perform descriptive analysis of demographic data and scores of symptoms severity of intermittent or persistent rhinitis (ie, nasal congestion, anterior or posterior rhinorrhea, sneezing and nasal itching). All results will be expressed as mean values standard deviation, or percentages in case of categorical variables. Symptoms improvement will be assessed using symptom severity scores registered (by physicians and patients) at the initial visit versus those recorded at the final visit. The contrast between means will be adjusted by recruitment centers (random factor), physicians' specialty (random factor), and demographic variables such as age, sex, body mass index (fixed factors in case of categories or covariates in case of continuous variables).

The frequency of adverse events will be recorded and in case of an important finding the investigators will search for risk factors using a nested sample from the same population and matched by age and sex.

ELIGIBILITY:
Inclusion Criteria:

1. All patients have to sign the informed consent or give verbal confirmation prior to their inclusion in the study.
2. Outpatient (external) male or female over 18 years and under 50 years.
3. Patients with active rhinitis (anterior or posterior rhinorrhea, sneezing, nasal congestion and itching) persistent (≥ 4 days a week for 4 consecutive weeks) or intermittent (< 4 days a week for ≤ 4 consecutive weeks).
4. Patient with medical history of rhinitis 2 years prior to their participation in this study and whose nasal symptoms have been severe enough to require continuous or intermittent treatment (it requires a patient's symptoms need treatment at least for a 4 weeks period).
5. Patient with the ability to understand the risks and benefits requirement while participating in the study and is able to accomplish the study treatment and with filling questionnaires and patient's diaries.

Exclusion Criteria:

1. Patient with other nasal disease including: nasal polyps or nasal trauma recent.
2. Patient with intranasal malformations (cysts and fistulas of the nose dorsum, prenasal space malformation, midline dystrophy, arrhinea, abnormalities of the tear ducts), or other conditions such as; recent nasal biopsy, drug rhinitis.
3. Non-controlled asthma or who were under systemic corticosteroid treatment.
4. Patient with Chronic Obstructive Pulmonary Disease.
5. Medical history of respiratory infection or other disease including bronchitis, pneumonia, common cold, acute or chronic sinusitis, influenza, etc. within 30 days prior to its inclusion in the study.
6. Patient receiving antibiotic therapy for any acute illness during the past 14 days.
7. Patient vaccinated against pneumococcus, H1N1 & seasonal influenza (past 30 days).
8. Patient required initiation or dose escalation immunotherapy. Immunotherapy is permitted if started 90 days ago and the patient received a stable dose during the last 30 days.
9. Patient has participated in another research study within 30 days preceding this visit.
10. Patient with medical history of hypersensitivity to steroids or any excipients of this class of drugs.
11. Treatment with systemic corticosteroids for a chronic or intermittent disorder (e.g., dermatitis) during the last six months or can present a condition that requires them.
12. Medical history of alcoholism and/or drug abuse in the last 2 years.
13. Medical history or positive testing for HIV, hepatitis B or C.
14. The patient uses any of drugs listed in the list on page 5 Table.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Male or female external patients over 18 years and under 50 years with active rhinitis (anterior or posterior rhinorrhea, sneezing, nasal congestion and itching) persistent (≥ 4 days a week for 4 consecutive weeks) or intermittent (<4 days a week for ≤ 4 consecutive weeks), with medical history of rhinitis 2 years prior to their participation in this study and whose nasal symptoms have been severe enough to require continuous or intermittent treatment (it requires a patient's symptoms need treatment at least for a 4 weeks period). All patients have to sign the informed consent or give verbal confirmation prior to their inclusion in the study.
Sampling Method: Non-Probability Sample
Enrollment: 1630 (Actual)
Dates: Start 2011-08; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Comparison symptoms´ score between initial score day 1 (V-0) vs. day 28 ± 2 (V-1). With a 7-point Likert scale. | 4 weeks
  The main outcome will be the described symptoms´ score and will be analyzed by comparison of the initial symptom score day 1 (V-0) vs. day 30 ± 2 (V-1). This is a quasi quantitative variable with a 7-point Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca AstraZeneca, Study Director — AstraZeneca
Locations (1):
- Yasmín Crespo, Naucalpan, State of Mexico, Mexico